CLINICAL TRIAL: NCT05212857
Title: Long-term Effects of Enhanced Systemic Therapy and Tumor-directed Therapy for Newly Diagnosed Oligometastatic Prostate Cancer Confirmed by Conventional Imaging Modality: a Prospective, Single-arm Study.
Brief Title: Enhanced Systemic Combined With Local Treatment for Primary and Metastatic Lesions in Oligo-metastatic Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMPCa-ENSURE
Record Dates: First submitted 2021-12-24; First posted 2022-01-28 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radical prostatectomy; androgen deprivation therapy; local treatment; radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; Goserelin; Triptorelin Pamoate; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Abiraterone Acetate; apalutamide; enzalutamide; Radiotherapy; Radiosurgery; Protons; Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- systemic treatment combined with radical treatment and radiotherapy (Experimental): All recruited participants would receive long-term and unified systemic treatment. Systemic treatment is defined as chemical castration plus new-generation anti-androgen therapy.
  For the primary lesion:
  The preferred local treatment for primary lesion is radical prostatectomy. Patients who refuse surgery or whose tumors cannot be surgically resected after 3 months' systemic treatment could receive radical radiotherapy.
  For the metastatic lesion:
  Radiotherapy for metastatic lesions would be performed between 4 weeks and 24 weeks after the local treatment for primary lesion. Stereotactic body radiation therapy (SBRT) is preferred, which could treat all the detected lesions at once or in stages.
  Interventions: Drug: Leuprolide acetate; Drug: Goserelin acetate; Drug: Triptorelin acetate; Drug: Degarelix acetate; Drug: Abiraterone acetate; Drug: Apalutamide; Drug: Enzalutamide; Procedure: Local treatment for primary lesion; Radiation: Radiotherapy for primary lesion; Radiation: Radiotherapy for metastatic lesion

INTERVENTIONS:
Drug: Leuprolide acetate — Given subcutaneously or as an injection
  Other Names: Enantone
Drug: Goserelin acetate — Given subcutaneously or as an injection
  Other Names: Zoladex
Drug: Triptorelin acetate — Given subcutaneously or as an injection
  Other Names: Diphereline
Drug: Degarelix acetate — Given subcutaneously or as an injection
  Other Names: Firmagon
Drug: Abiraterone acetate — Given orally
  Other Names: ZYTIGA
Drug: Apalutamide — Given orally
  Other Names: ERLEADA
Drug: Enzalutamide — Given orally
  Other Names: Xtandi
Procedure: Local treatment for primary lesion — Radical prostatectomy to remove prostate primary lesion
Radiation: Radiotherapy for primary lesion — Radical radiotherapy for primary lesion
Radiation: Radiotherapy for metastatic lesion — Stereotactic body radiation therapy or proton and heavy ion radiation therapy is preferred, which could treat all the lesions at once or treat different lesions in stages.
  Other Names: Stereotactic body radiation therapy or proton and heavy ion radiation therapy

SUMMARY:
Oligo-metastatic prostate cancer (OMPCa) is considered as an intermediated state between localized and poly-metastatic disease. Various retrospective studies and prospective clinical trials are carrying out to validate whether patients with OMPCa could benefit from local treatment for both primary and metastatic lesions. The investigators here to conduct a unique clinical trial which OMPCa patients were confirmed by conventional imaging, and received a long-term enhanced systemic therapy accompanied by tumor-directed therapy.

DETAILED DESCRIPTION:
Recent studies showed that metastatic lesion of prostate cancer may originate from both the primary and the existing metastatic lesion, thus, disease with limited number of metastatic lesions were considered as oligo-metastatic prostate cancer (OMPCa), an intermediated state between localized and poly-metastatic disease. For patients with newly diagnosed OMPCa, serval studies revealed that prostate radiation therapy could improve their clinical outcomes. For patients with oligo-recurrent prostate cancer, they could also be benefit from stereotactic ablative radiation therapy to the metastatic lesion. The investigators thus designed a distinct clinical trial including patients who were confirmed as oligo-metastatic disease by conventional imaging modality (CT, MRI and ECT) rather than PSMA PET-CT. This study also aimed to evaluate the therapeutic effects of tumor-directed treatment under the background of long-term enhanced systemic therapy, including abiraterone, enzalutamide or apalutamide. Here, the investigators proposed that, for patients with de novo oligo-metastatic prostate cancer, enhanced systemic treatment combined with radical treatment of primary lesion and radiotherapy of all accessible metastatic lesions may prolong their survival time without affecting their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed de novo prostate adenocarcinoma (can be accompanied by neuroendocrine differentiation, but accounts for less than 10% of the total tumor components);
2. Aged between 18 and 80;
3. M1a/b disease with presence of 1-5 visible metastases (detected by bone scan (ECT), chest, abdominal and pelvic CT or MRI). Biopsy of the suspected metastases is recommended to the patients. If the patients refused to the biopsy, additional PSMA-PET/CT or regional MRI should be performed to confirm the metastatic lesions.
4. The metastatic lesions should meet the following the criteria:

   1. Metastases are limited to bone or lymph nodes;
   2. Visceral metastases are not allowed;
   3. Radiographic observed pelvic lymph node metastasis with a diameter of >2cm should also be considered as one metastatic lesion.
   4. If the lymph nodes are the only detected metastatic lesions, at least one metastatic lymph node should be outside the pelvis.
5. ECOG performance status of 0 or 1;
6. PSA less than 100ng/ml at diagnosis;
7. No more than one month's systemic treatment before enrollment (including castration (surgical or medical castration), castration combined with traditional anti-androgen therapy (flutamide or bicalutamide));
8. No previous pelvic radiotherapy history;
9. The primary lesion of prostate cancer has not received any form of local treatment (surgery, radiotherapy, cryotherapy, radiofrequency ablation, etc.); TURP is allowed, if the aim of the surgery is to relieve lower urinary tract symptom but not to treat the tumor.
10. The metastatic lesions of prostate cancer have not received any form of local treatment (surgery, radiotherapy, cryotherapy, radiofrequency ablation, etc.);
11. Written informed consent;
12. Willing and expected to comply with treatment and follow up schedule.
13. Life expectancy > 10 years.

Exclusion Criteria:

1. Received prior local treatment for primary lesion or metastatic lesions, including radical prostatectomy, radical radiotherapy, surgery or radiotherapy to metastatic lesion;
2. Received prior systemic treatment for prostate cancer longer than 1 month;
3. Received prior castration combined with new-generation androgen signaling pathway inhibitors such as abiraterone, apalutamide or enzalutamide; castration combined with docetaxel chemotherapy;
4. Had any visceral metastases (liver, lung, brain etc.);
5. Histologically or cytologically confirmed small cell carcinoma;
6. Unable to tolerate the treatment for primary and metastatic lesion;
7. Unwilling to accept potential related adverse events caused by treatment for primary and metastatic lesion;
8. Had any other previous or current malignant disease, except for curatively treated skin basal cell carcinoma or other tumors cured for more than 5 years;
9. Had other severe disorders, such as:

   1. Unstable cardiac disease,
   2. Myocardial infarction less than 6 months prior to enrollment,
   3. Clinically significant cardiac failure requiring treatment, defined as New York Heart Association (NYHA) class III,
   4. Uncontrolled hypertension,
   5. Severe neurological or psychological disorder including dementia or epilepsy,
   6. Uncontrolled active infection,
   7. Acute gastric ulcer,
   8. Hypercalcemia,
   9. Chronic obstructive pulmonary lung disease requiring hospitalization,
   10. Any other significant disorders that in the investigator's opinion means the participant is unfit for any of the study treatments;
10. Had participated in other clinical trial before enrollment.
11. Had contraindications to radiotherapy or unsuitable for radical radiotherapy evaluated by radiologists and physicists.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Two years' radiographic progression-free survival (rPFS) | 2 years
  Proportion of patients without radiographic progression after two years' treatment.
  The soft-tissue lesion evaluation criterion was RECIST1.1, and the bone lesion evaluation criterion was PCWG3

SECONDARY OUTCOMES:
Two years' overall survival (OS) | 2 years
  Proportion of patients survived after two years' treatment.
Two years' PSA progression-free survival (PSA-PFS) | 2 years
  Proportion of patients with no observed PSA progression after two years' treatment. PSA progression is defined as a confirmed increase in the PSA level from the nadir value by ≥25% and by ≥2 ng/ml.
Pathological complete response (pCR) or minimal residual disease (MRD) rate | 1 month after prostatectomy as local treatment for primary lesion.
  Pathological response, defined as achieving either pCR or MRD at radical prostatectomy (RP). pCR is defined as the absence of morphologically identifiable carcinoma in the RP specimen. MRD will be defined as residual tumor in the RP specimen measuring ≤ 5 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Doctoral, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No